CLINICAL TRIAL: NCT05911711
Title: Identification and Clinical Efficacy Analysis of Biomarkers in Sepsis Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kangdong Sacred Heart Hospital (Other)
Collaborators: Chungnam National University (Other); Chungnam National University Hospital (Other)
Responsible Party: Principal Investigator, So Young Park, associate professor, Kangdong Sacred Heart Hospital
Other Study IDs: 2022-03-015-004
Record Dates: First submitted 2023-06-07; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Biospecimen Retention: Samples Without DNA — Blood for (RNAseq) Bronchoalveolar lavage (for microbiome)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sepsis patient in Medical ICU: Eligibility Criteria:
  adults over the age of 19 a sepsis patient in Medical ICU
  Patients are excluded from the study :
  If the patient or care giver does not agree to participate in the study a bone marrow transplant or an organ transplant patient a Do not resuscitation (DNR) patient
  Interventions: Other: Prognostic factor

INTERVENTIONS:
Other: Prognostic factor — normal person (no sepsis group)

SUMMARY:
Sepsis, a severe response to bacterial infection, lacks understanding of immunometabolic features that can identify high-risk patients. This study aimed to discover immune, biological, and metabolic biomarkers in sepsis patients with poor prognosis and understand the underlying mechanisms of host immune responses.

DETAILED DESCRIPTION:
Sepsis is a life-threatening condition resulting from a dysregulated host response to infection and remains a significant global health crisis. Accurately identifying high-risk patients and understanding the underlying mechanisms of distinct host responses are crucial. Dysregulation of immune and biological responses, along with metabolic remodeling, has emerged as a prevalent characteristic in sepsis patients. However, there is still a need for a comprehensive understanding of specific markers related to immunometabolism and the underlying mechanisms contributing to the disturbance in sepsis pathogenesis.

This study aims to investigate the immune, biological, and metabolic profiles of sepsis patients, focusing on the alteration of metabolism in sepsis patients with poor outcomes. The findings of this study will provide valuable insights into dysregulated immunometabolism, shedding light on its contribution to the potentiation of immunopathogenesis in sepsis.

Eligibility Criteria adults over the age of 19 a sepsis patient in ICU

Patients are excluded from the study If the patient or care giver does not agree to participate in the study a bone marrow transplant or an organ transplant patient a Do not resuscitation(DNR) patient a patient under the age of 18

Outcome Measure ICU mortality, 28 days mortality Use of inotropics, vasopressors CRRT(continuous renal replacement therapy), ECMO (Extracorporeal membrane oxygenation), Interventional lung assist, polymyxin

ELIGIBILITY:
Inclusion Criteria:

* adults over the age of 19 a sepsis patient in ICU

Exclusion Criteria:

* If the patient or care giver does not agree to participate in the study a bone marrow transplant or an organ transplant patient a DNR patient a patient under the age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: sepsis patient in Medical ICU sepsis definition : Sepsis is life-threatening organ dysfunction caused by a dysregulated host response to infection
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-07-07 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-06-07 (Estimated)

PRIMARY OUTCOMES:
up to 1 day ICU mortality" | up to 1 day ICU mortality"
  up to 1 day ICU mortality"

SECONDARY OUTCOMES:
28 days mortality | 28 days mortality
  28 days mortality

CONTACTS AND LOCATIONS:
Overall Officials: So Young Park, doctor, Study Chair — Kangdong Sacred Heart Hospital
Locations (1):
- KangdonSHH, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
This study complies with the Helsinki Declaration, is conducted in accordance with the test plan approved by the Institutional Bioethics Committee (IRB) of Kangdong Sacred Heart Hospital, and will be conducted in accordance with the clinical trial management standards (GCP) set by the Korea Food and Drug Administration. Personal information is not included in the research results, and for this purpose, personal information will not be included even when the research results are published and the research results are disclosed by assigning a code number to the research results. Clinical Information Analysis reviews patient's charts and the lead researcher is responsible for the supervision of the state to ensure that personal information collected before being coded is not leaked.
Supporting Information: ICF
Time Frame: Keeping research-related records for three years from the time the research is completed pursuant to Article 15 of the Enforcement Rule of the Bioethics and Safety Act
Access Criteria: adults over the age of 19 a sepsis patient in Medical ICU

REFERENCES:
- [Background] Park SY, Shrestha S, Youn YJ, Kim JK, Kim SY, Kim HJ, Park SH, Ahn WG, Kim S, Lee MG, Jung KS, Park YB, Mo EK, Ko Y, Lee SY, Koh Y, Park MJ, Song DK, Hong CW. Autophagy Primes Neutrophils for Neutrophil Extracellular Trap Formation during Sepsis. Am J Respir Crit Care Med. 2017 Sep 1;196(5):577-589. doi: 10.1164/rccm.201603-0596OC. PMID 28358992
- [Derived] Roh T, Ju S, Park SY, Ahn Y, Chung J, Nakano M, Ryu G, Kim YJ, Kim G, Choi H, Lee SG, Kim IS, Lee SI, Chung C, Shimizu T, Miyoshi E, Jung SS, Park C, Yamasaki S, Park SY, Jo EK. Fucosylated haptoglobin promotes inflammation via Mincle in sepsis: an observational study. Nat Commun. 2025 Feb 4;16(1):1342. doi: 10.1038/s41467-025-56524-3. PMID 39904983